CLINICAL TRIAL: NCT03561844
Title: Investigate the Efficacy and Effectiveness of Aromatherapy for the Management of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, professor and head of rehabilitation science department, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P17-0203-2
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aromatherapy-scent (Active Comparator)
  Interventions: Other: aromatherapy
- aromatherapy-touch (Active Comparator)
  Interventions: Other: aromatherapy
- waiting-list control (No Intervention)

INTERVENTIONS:
Other: aromatherapy — Each of participants in the aromatherapy (inhalation) group will receive inhalation aromatherapy and those in the aromatherapy (massage) group will receive aromatherapeutic massage. As to the waiting control group, participants will be given either one of these two interventions after the implementation phase is completed.
  Arms: aromatherapy-scent; aromatherapy-touch

SUMMARY:
In recent decades, following an increased longevity in Hong Kong, there is a drastic increase in the prevalence chronic conditions, including chronic pain, seems to be the main reasons of suffering for many older adults. This condition not only pose a burden to the whole family but also the healthcare system.

While conventional treatment of chronic pain using pharmacotherapy and non-pharmacological treatments has been effective for managing symptoms, owing to the adverse side effects caused by anti-psychotic drugs and the short effective period incurred by non-pharmacological interventions, development of alternative and non-pharmacological approaches for the management of pain is of urgent need. Research has shown that aromatherapy (both administered through inhalation and therapeutic massage) has been effective in reducing showing pain-relieving effects. These findings support the premise that aromatherapy and the investigators hope to provide further evidence to support the use of aromatherapy as an evidence-based mainstream intervention for pain relief in older adults with chronic pain.

Whilst there is sufficient evidence to support the effectiveness of aromatherapy, few studies compared the effectiveness of the use of aromatherapy by inhalation and/or therapeutic massage. The investigators aim to address the above research gaps on the clinical application of aromatherapy on chronic pain, with a focus on comparing the differential effectiveness between administration by inhalation and administration by therapeutic massage. The proposed research aims to (1) test the efficacy and effectiveness of aromatherapy on the symptom management of chronic pain in older adults; (2) compare the effects of aromatherapy-scent (i.e., inhalation) and aromatherapy-touch (i.e., therapeutic massage) in older adults with chronic pain. This study also explores the benefits of aromatherapy on cognitive functioning, functional performance and social engagement as secondary outcomes.

A randomized, controlled, and single blinded trial is proposed. 120 older adults with chronic pain will be randomly assigned to aroma inhalation (intervention), aroma-touch or wait-list (control) treatments. Pain intensity and subjective changes in mood states (primary outcome), cognitive functioning, functional performance and social engagement (secondary outcome) will be assessed three times: pre-treatment, mid-treatment, post-treatment. If the study hypotheses are supported, the findings will provide empirical support for a treatment option that could improve manage the symptoms of patients diagnosed with chronic conditions, and also improve cognitive functioning, functional performance, and social engagement of older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* having a CMMSE score over or equal to 15
* having chronic pain or a widespread pain condition such as fibromyalgia for at least 3 months
* be willing to participate in the research, with informed consent signed by their guardian or carer.

Exclusion Criteria:

* being allergic to essential oils
* refusal to give consent
* being over-sensitive to tactile stimulation
* having a history of kidney and liver disease
* no history of an epileptic seizure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | the change from baseline to the completion of intervention (16 weeks later)
  Numerical Rating Scale (NRS) will be used to measure the changes of pain among three time points within four months. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Cantonese Version of the Mini-mental State Examination (CMMSE) | baseline, 8 weeks after baseline, and 16 weeks after baseline
  Cantonese Version of Mini-mental State Examination (MMSE) is a brief 30-point questionnaire used to assess the change of the cognitive functions among three time points at four months. The range of the score is from 0 point to 30 points, which a lower score indicates the worse cognitive functions.
Chinese Version of the Barthel Index-100 | baseline, 8 weeks after baseline, and 16 weeks after baseline
  Chinese Version of the Barthel Index-100 is used to measure the change of the performance in activities of daily living (ADL) among three time points at four months. Scores range from 0 to 100, with higher scores indicating greater independence.
Index of Social Engagement(ISE) | baseline, 8 weeks after baseline, and 16 weeks after baseline
  The change of the social engagement among three time points at four months will be measured using the 6-item index of social engagement (ISE). Total scores on the ISE can range from 0 to 6, with a higher score indicating a higher level of social engagement.
Profile of Mood States (POMS)- Shorterned Chinese Version | baseline, 8 weeks after baseline, and 16 weeks after baseline
  The Chinese abbreviated version of the Profile of Mood States will be used to subjective changes in mood states among three time points at four months. There are 40 items, where participants will rate on a scale of 0(not at all)-5(extremely) and higher score indicates more distress.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No